CLINICAL TRIAL: NCT00989040
Title: Impact of Neuropathic Post-zosterian Pain on the Cognition (NPZ and Cognition)
Brief Title: Impact of Neuropathic Post-Zosterian Pain on the Cognition
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0049
Record Dates: First submitted 2009-03-13; First posted 2009-10-02 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Neuropathic Post-zosterian Pain; Cognition
Keywords: NPZ; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

INTERVENTIONS:
Drug: usual treatment: Versatis — * To explore if the cognition is failed in treated patients suffering of neuropathic postzosteria pain.
  * To see if treated patients with patch (Versatis®) have better cognition than treated patients without patch.

SUMMARY:
Pain is defined as a sensorial and emotional phenomenon and lead consequences on the cognition. These consequences could be increased with usual treatment. So the aim of this study is to explore these cognitive consequences.

DETAILED DESCRIPTION:
Pilot prospective study with parallel groups

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering of NPZ pain
* Over 55 years old
* Healthy volunteers

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who suffer of neuropathic post-zosteria pain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The principal outcome is to explore if the cognition is failed in treated patients suffering of neuropathic post-zosteria pain. | at day 1

SECONDARY OUTCOMES:
Study if treated patients with patch (Versatis®) have better cognition than treated patients without patch. | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Claude Dubray, PUPH, Principal Investigator — CIC-CPC Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Pickering G, Pereira B, Clere F, Sorel M, de Montgazon G, Navez M, Picard P, Roux D, Morel V, Salimani R, Adda M, Legout V, Dubray C. Cognitive function in older patients with postherpetic neuralgia. Pain Pract. 2014 Jan;14(1):E1-7. doi: 10.1111/papr.12079. Epub 2013 May 23. PMID 23701810